CLINICAL TRIAL: NCT06550921
Title: Ablation of Oligometastasis Combined With Lenvatinib and PD-1 Inhibitor for Advanced Hepatocellular Carcinoma: A Multicenter, Prospective, Phase II Study
Brief Title: Ablation of Oligometastasis Combined With Lenvatinib and PD-1 Inhibitor for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 8
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Advanced Hepatocellular Carcinoma; Oligometastasis; Ablation; Anti-PD1 Antibody; Lenvatinib
Keywords: Lenvatinb; Tislelizumab; Sintilimab; Camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation-Len-PD-1 inhibitor (Experimental): ablation of oligometastasis therapy combined with lenvatinib and PD-1 inhibitor
  Interventions: Procedure: ablation of oligometastasis

INTERVENTIONS:
Procedure: ablation of oligometastasis — The oligometastasis of hepatocellular carcinoma are ablation completely by ablation (including microwave ablation, radiofrequency ablation, and cryoablation)

SUMMARY:
Ablation has been an effective approach for treating intrathoracic metastases. However, for hepatocellular carcinoma with oligometastasis, ablation of metastases remains relatively unexplored.

DETAILED DESCRIPTION:
Systemic therapy is the standard treatment for advanced hepatocellular carcinoma (HCC) with metastasis. However, metastases with limited number (oligometastasis) can represent a subtype and transition point between localized disease and widespread metastases. Thus, eliminating metastases could be advantageous and beneficial to the prognosis if feasible and permitted. Image-guided ablation therapy, such as microwave ablation (MWA), radiofrequency ablation (RFA), and cryoablation, has attracted great interest as a minimally invasive approach against intrathoracic metastases. Recently, ablation has been used on patients with pulmonary metastases from various cancers. This technique yields high proportions of sustained complete responses and is associated with relatively low morbidity. Thus, we conduct this multicenter single arm study to explore the efficacy, safety of lenvatinib and PD-1 inhibitor with metastases-directed ablation in advanced HCC. This study focuses on the management of ablation of oligometastasis therapy combined with lenvatinib and PD-1 inhibitor. This study aims to evaluate the survival benefits of ablating oligometastasis for advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of primary HCC, confirmed histologically or clinically according to the criteria of the American Association for the Study of Liver Diseases 20;
2. presence of oligometastasis, the metastases found within three month of HCC diagnosis;
3. metastases with limited five sites and no more two organs involved, with a maximum diameter of ≤5cm;
4. receipt of Lenvatinib and PD-1 inhibitor as the first-line systemic therapy for a minimum of 3 months before study ablation, with controlled intrahepatic tumors and no progression of metastases. Controlled intrahepatic tumors were defined as those showing a partial or stable response according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST);
5. undergone locoregional treatments, including transarterial artery chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC);
6. classified as Child-Pugh class A or B and having an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. no history of other malignancies.
8. life expectancy more than 3 months;
9. agreed to participated in this clinical trial;
10. Hemameba ≥3.0 x109/L, neutrophil ≥1.5x109/L, hemoglobin≥10.0 g/L, platelet≥100x 109/L, ALT; AST; bilirubin ≤1.5-fold normal, GFR≥60ml/min.

Exclusion Criteria:

1. recurrent HCC;
2. advanced HCC Lenvatinib and PD-1 inhibitor treated with as second systemic therapy;
3. age < 18 years or > 75 years;
4. advanced HCC with more than five metastases;
5. no response to Lenvatinib;
6. metastases size > 5 cm;
7. life expectancy less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | 24 months
  Progression-Free-Survival (PFS)

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.
Adverse events | 24 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: No